CLINICAL TRIAL: NCT05766475
Title: Group-based Prevention of Postpartum Depression: In-person vs. Virtual Delivery
Brief Title: In-person vs. Virtual Delivery of a Group-based Prevention of Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Denver Health Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1916994-3; R01MH130976-01 (NIH)
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Depression
Keywords: Prenatal depression; health disparities; preventative intervention; virtual therapy; interpersonal therapy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Delivery of Group Preventative Intervention (ROSE) (Active Comparator): The Reach Out, Stay Strong, Essentials for New Mothers Program (ROSE), is an established Interpersonal Therapy (IPT)-oriented group intervention for postpartum depression. ROSE is a brief (5-session) program and its content addresses social support, role transition to motherhood, communication skills, and psychoeducation on PPD. ROSE consists of four 90-minute, weekly in person group sessions and one individual booster session. The first four sessions of ROSE will be delivered in groups of 6 to 20, and conducted in both English and Spanish. For the in-person groups, transportation via Uber will be provided to Denver Health Medical Center to reduce barriers to attendance.
  Interventions: Behavioral: ROSE Program: In Person
- Virtual Delivery of Group Preventative Intervention (ROSE) (Experimental): In parallel to ROSE delivered in person, virtual ROSE consists of four 90-minute, weekly group sessions conducted via Zoom and one individual booster session.
  Interventions: Behavioral: ROSE Program: Virtual

INTERVENTIONS:
Behavioral: ROSE Program: In Person — In-person preventative intervention for postpartum depression that includes content on building social support and communication skills in relationships, navigating the role transition to motherhood, and learning about signs and symptoms of depression after delivery.
  Other Names: Rose; Group IPT; La Luz
  Arms: In-Person Delivery of Group Preventative Intervention (ROSE)
Behavioral: ROSE Program: Virtual — Virtual ROSE covers the same content (e.g. improving social support and communication) and is delivered by the same facilitators as the in-person intervention via telehealth.
  Arms: Virtual Delivery of Group Preventative Intervention (ROSE)

SUMMARY:
The goal of this clinical trial is to test whether an established preventive intervention (group interpersonal therapy) delivered virtually shows the same benefits for preventing postpartum depression as it does when delivered in person.

DETAILED DESCRIPTION:
Depression is one of the most common perinatal complications, with 1 in 7 mothers qualifying for a diagnosis of postpartum depression (PPD) and even higher rates for those who identify as Hispanic/Latine, Black or African American, American Indian, or Alaska Native, or by multiple races or ethnicities. This project addresses this major gap in services to prevent PPD, particularly among socioeconomically disadvantaged and minoritized groups. It tests the benefit of a virtual perinatal preventive intervention in English and Spanish to increase access, scalability and address the mental health needs of underserved populations. This project will test the virtual version against the in-person version of a service-ready efficacious preventive intervention in a randomized controlled trial (RCT). This trial will provide a test of a preventive intervention with a strong evidence base that is scalable and can be delivered with fidelity by service providers in settings where obstetric care is received. In this project, pregnant women will be randomized to receive an evidence-based group prevention program (Reach Out, Stay Strong, Essentials for New Moms; ROSE) designed for perinatal populations either a) in person, delivered at the hospital where they are receiving prenatal care or b) virtually, delivered by the same staff via video conferencing, both offered in English and Spanish. Diverse pregnant individuals (N = 900) will be randomized to receive virtual or in-person ROSE. The central outcome, depression, will be assessed via REDCap surveys, prenatally (before the program begins and at the end of gestation) and postpartum (approximately six-weeks, 3, 6, and 12-months after birth). Electronic health records (EHRs) and surveys will be used to examine obstetric, mental health (e.g., standard of care depression screening), and sociodemographic factors linked to health disparities that may impact who benefits most.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Less than 30 gestational weeks

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Symptom Checklist 20 (SCL 20) | 6 weeks after birth
  Self reported depression scores. Possible range of scores is 0 to 80, with the higher scores indicating higher depression levels.
Symptom Checklist 20 (SCL 20) | 3 months after birth
  Self reported depression scores.Possible range of scores is 0 to 80, with the higher scores indicating higher depression levels.
Symptom Checklist 20 (SCL 20) | 6 months after birth
  Self reported depression scores
Symptom Checklist 20 (SCL 20) | 12 months after birth
  Self reported depression scores. Possible range of scores is 0 to 80, with the higher scores indicating higher depression levels.
Center for Epidemiologic Studies Depression Scale (CES-D) | 6 weeks after birth
  Self reported depression scores. Possible range of scores is 0 to 60, with the higher scores indicating higher depression levels.
Center for Epidemiologic Studies Depression Scale (CES-D) | 3 months after birth
  Self reported depression scores. Possible range of scores is 0 to 60, with the higher scores indicating higher depression levels.
Center for Epidemiologic Studies Depression Scale (CES-D) | 6 months after birth
  Self reported depression scores. Possible range of scores is 0 to 60, with the higher scores indicating higher depression levels.
Center for Epidemiologic Studies Depression Scale (CES-D) | 12 months after birth
  Self reported depression scores. Possible range of scores is 0 to 60, with the higher scores indicating higher depression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Galena Rhoades, PhD, Principal Investigator — University of Denver; Elysia P Davis, PhD, Principal Investigator — University of Denver
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared in accordance with NIMH Data Archive requirements.

REFERENCES:
- [Derived] Liu DY, Perry NS, Demers CH, Hyer JS, Alamo A, Vuksanovich P, Dube N, Flanagan ER, Gallop RJ, Rhoades GK, Davis EP. Virtual versus in-person ROSE program (La Luz) as universal prevention for perinatal depression: Protocol for a randomized controlled trial in a safety net hospital. Contemp Clin Trials. 2025 Aug;155:107988. doi: 10.1016/j.cct.2025.107988. Epub 2025 Jun 15. PMID 40527396